CLINICAL TRIAL: NCT06656065
Title: Index Microvascular Resistance (IMR) in Heart Transplant Patients
Brief Title: IMR-Heart Trasplant Study
Status: Recruiting | Type: Observational
Sponsor: Hospital Miguel Servet (Other)
Collaborators: Central University Hospital of Asturias (Unknown); University Hospital La Fe, Valencia (Unknown); University Hospital Virgen de la Arrixaca, Murcia (Unknown); University Hospital 12 Octubre, Madrid (Unknown); University Hospital Reina Sofia, Cordoba (Unknown); Bellvitge University Hospital (Unknown); University Hospital Virgen del Rocio, Sevilla (Unknown)
Responsible Party: Principal Investigator, Georgina Fuertes Ferre, Dr. Fuertes, Hospital Miguel Servet
Other Study IDs: C.I. PI23/242
Record Dates: First submitted 2024-10-15; First posted 2024-10-24 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Heart Transplant Rejection; Microvascular Resistance
Keywords: Heart Trasplant; Acute cellular rejection; IMR; Endomyocardial biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IMR≥15: Heart trasplant patient with an index of microvascular resistance ≥ 15 measured in the first three months in the physiological study.
- IMR<15: Heart trasplant patient with an index of microvascular resistance<15 measured in the first three months in the physiological study.

SUMMARY:
Acute allograft rejection (AAR) is an important cause of morbi-mortality in heart transplant (HT) patients, particularly during the first year. Endomyocardial biopsy (EMB) is the "gold standard" to guide post- heart transplantation treatment. However, it is associated with complications that can be potentially serious. The index of microvascular resistance (IMR) is a specific physiological parameter used to assess microvascular function. Invasive coronary assessment has been shown to be both feasible and safe. Detection of coronary microvascular dysfunction (MCD) by IMR may help to identify high risk HT patients. In fact, an increased IMR measured early after HT has been associated with AAR, higher all-cause mortality and adverse cardiac events. A high IMR value early after HT may identify patients at higher risk who require increased surveillance or adjustments in immunosuppressive therapy. Conversely, a low IMR value may support reducing the number of EMBs. Our aim is to evaluate IMR in heart transplant patients within the first year. Changes in management after knowing IMR values and prognostic implications of IMR in a long term follow up will also be assessed.

DETAILED DESCRIPTION:
The IMR-HT study is a multicenter, prospective observational study that will include post-HT stable patients undergoing coronary physiological assessment in the first three months and one year.

Assessment of IMR, coronary flow reserve (CFR) and fractional flow reserve (FFR) will be performed using the standard thermodilution technique. The left anterior descending coronary artery will be evaluated in all patients. Circumflex or right coronary artery could be additionally evaluated at operator's discretion. An intracoronary pressure and temperature sensor-tipped guidewire (Pressure Wire TM X guide- wire 0.014', Abbott, IL, USA) will be used to perform the measurements. The tip pressure sensor will be advanced into the mid-to-distal portion of the evaluated vessel. Baseline aortic pressure (Pa) and distal intracoronary pressure (Pd) will be obtained to calculate the resting index Pd/Pa. To measure the mean transit time (Tmn) under basal conditions, intracoronary administration of 3 mL of room-temperature saline will be manually injected three times in succession (3 mL/s). Then maximal hyperemia will be induced using adenosine iv (140 to 180 mg/kg/min) and three additional intracoronary room temperature saline boluses of 3 ml will be administered to determine the mean transit time at hyperemia (Tmnh). Finally, fractional flow reserve (FFR), coronary flow reserve (CFR) and IMR will be calculated using the software Coroventis Coroflow (Coroventis Abbott, Uppsala, Sweden).

Changes in HT patient management (number of EMBs, immunosuppressive therapy modifications) after knowing IMR values will also be assessed.

Based on previously published clinical data on IMR in heart transplant patients, a post-HT management algorithm is proposed:

* IMR < 15: The frequency of biopsies could be reduced or maintained as per protocol. No changes to immunosuppressive therapy would be required.
* IMR ≥ 15: Biopsies would be performed at the standard frequency according to protocol. Immunosuppressive therapy could be intensified or maintained the same.

Of note, given the observational characteristics of the study, clinical management decisions will be made at the discretion of the treating physician, taking into account the patient's clinical condition and other complementary tests.

Both groups (IMR<15 vs IMR≥15) will be compared in terms of cardiac events occurrence.

Clinical conditions, laboratory findings and clinical events will be assessed at one month and one year. Follow up will be extended for up to five years. Data will be included in an online database specifically designed for the study on platform REDCap (Research Electronic Data Capture).

A number will be assigned to each patient; their identity will not be disclosed in any case. All shared information will be anonymized. The principal investigator at each center will be responsible for keeping the data anonymized.Data will be processed in accordance with the protection legislation in force (Spanish Personal Data Protection and Guarantee of Digital Rights Act 3/2018, and Regulation (EU) 2016/679).

Our aim will be to assess IMR values in heart transplant patients within one year and evaluate changes in management after knowing of IMR values. We believe it is important to move forward in AAR surveillance and reduce the number of endomyocardial biopsies. In addition to assessing their diagnostic capabilities, IMR should also be assessed based on clinical outcomes. Therefore, we are convinced the results of this trial will be very important for our HT patient population.

ELIGIBILITY:
Inclusion Criteria:

* Heart transplant patients >18 years.
* Patients who have received and signed informed consent.

Exclusion Criteria:

* Patients with hemodynamic instability after HT, including cardiogenic shock or severe coagulopathy.
* Patients with acute cellular rejection before intracoronary physiological assessment.
* Patients with bronchial asthma or bronchopathy with a positive bronchodilation test, which contraindicates the use of adenosine.
* Patients with epicardial coronary lesions with a resting physiological index ≤0.89 or ≤0.80 at hyperemia.
* Patients unlikely to cooperate or with inability or unwillingness to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart trasplant patients that have signed informed consent and meet all inclusion and exclusion criteria for undergoing IMR assessment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2028-05-23 (Estimated); Study Completion 2028-10-14 (Estimated)

PRIMARY OUTCOMES:
IMR values in the first three months and one year after heart transplant | One year
  IMR measured by the invasive thermodilution technique. IMR is defined as the distal coronary pressure divided by the inverse of the hyperemic mean transit time and is expressed in units of mmHg.s.

SECONDARY OUTCOMES:
IMR variation between first three months after HT and one year | One year
  Comparison between the values of index of microvascular resistance (IMR) measured by bolus thermodilution technique between the first and 3rd month after HT and one year in the invasive physiological study. IMR may be expressed as mmHg·s.
Acute cellular rejection | One year
  A ≥2R degree according to the 2010 ISHLT system. Two or more focal infiltration points associated with myocyte injury in EMB. Diffuse infiltration with multi-focal myocyte injury with/without oedema, hemorrhage or vasculitis.
Cardiac allograft vasculopathy | Five years
  Accelerated fibroproliferative process characterized by diffuse, concentric and longitudinal thickening of the intima of the vascular tree of the graft, affecting everything from the major epicardial arteries to the coronary microvasculature.
Cardiovascular mortality | Five years
  Caused by cardiovascular disease or unknown death
Heart failure | Five years
  Diastolic or systolic heart failure after heart transplant
Inmunosupressive therapy | Five years
  Changes in any of the inmunosuppresive agents pre-established in each center heart transplant protocol
EMB performed in each center within the first year | One year
  The number of biopsies performed by each center, after knowing IMR baseline values.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Miguel Servet, Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP
Time Frame: October 2024
Access Criteria: All researches/physicians involved in this investigational field

REFERENCES:
- [Background] Lee JM, Choi KH, Choi JO, Shin D, Park Y, Kim J, Lee SH, Kim D, Yang JH, Cho YH, Sung K, Choi JY, Park M, Kim JS, Park TK, Song YB, Hahn JY, Choi SH, Gwon HC, Oh JK, Jeon ES. Coronary Microcirculatory Dysfunction and Acute Cellular Rejection After Heart Transplantation. Circulation. 2021 Nov 2;144(18):1459-1472. doi: 10.1161/CIRCULATIONAHA.121.056158. Epub 2021 Sep 3. PMID 34474597
- [Background] Okada K, Honda Y, Luikart H, Yock PG, Fitzgerald PJ, Yeung AC, Valantine HA, Khush KK, Fearon WF. Early invasive assessment of the coronary microcirculation predicts subsequent acute rejection after heart transplantation. Int J Cardiol. 2019 Sep 1;290:27-32. doi: 10.1016/j.ijcard.2019.04.018. Epub 2019 Apr 8. PMID 30987835
- [Background] Ahn JM, Zimmermann FM, Gullestad L, Angeras O, Karason K, Russell K, Lunde K, Okada K, Luikart H, Khush KK, Honda Y, Pijls NHJ, Lee SE, Kim JJ, Park SJ, Solberg OG, Fearon WF. Microcirculatory Resistance Predicts Allograft Rejection and Cardiac Events After Heart Transplantation. J Am Coll Cardiol. 2021 Dec 14;78(24):2425-2435. doi: 10.1016/j.jacc.2021.10.009. PMID 34886963
- [Background] Hiemann NE, Wellnhofer E, Knosalla C, Lehmkuhl HB, Stein J, Hetzer R, Meyer R. Prognostic impact of microvasculopathy on survival after heart transplantation: evidence from 9713 endomyocardial biopsies. Circulation. 2007 Sep 11;116(11):1274-82. doi: 10.1161/CIRCULATIONAHA.106.647149. Epub 2007 Aug 20. PMID 17709643
- [Background] Saraiva F, Matos V, Goncalves L, Antunes M, Providencia LA. Complications of endomyocardial biopsy in heart transplant patients: a retrospective study of 2117 consecutive procedures. Transplant Proc. 2011 Jun;43(5):1908-12. doi: 10.1016/j.transproceed.2011.03.010. PMID 21693299
- [Background] Khush KK, Cherikh WS, Chambers DC, Harhay MO, Hayes D Jr, Hsich E, Meiser B, Potena L, Robinson A, Rossano JW, Sadavarte A, Singh TP, Zuckermann A, Stehlik J; International Society for Heart and Lung Transplantation. The International Thoracic Organ Transplant Registry of the International Society for Heart and Lung Transplantation: Thirty-sixth adult heart transplantation report - 2019; focus theme: Donor and recipient size match. J Heart Lung Transplant. 2019 Oct;38(10):1056-1066. doi: 10.1016/j.healun.2019.08.004. Epub 2019 Aug 10. No abstract available. PMID 31548031
- [Background] Costanzo MR, Dipchand A, Starling R, Anderson A, Chan M, Desai S, Fedson S, Fisher P, Gonzales-Stawinski G, Martinelli L, McGiffin D, Smith J, Taylor D, Meiser B, Webber S, Baran D, Carboni M, Dengler T, Feldman D, Frigerio M, Kfoury A, Kim D, Kobashigawa J, Shullo M, Stehlik J, Teuteberg J, Uber P, Zuckermann A, Hunt S, Burch M, Bhat G, Canter C, Chinnock R, Crespo-Leiro M, Delgado R, Dobbels F, Grady K, Kao W, Lamour J, Parry G, Patel J, Pini D, Towbin J, Wolfel G, Delgado D, Eisen H, Goldberg L, Hosenpud J, Johnson M, Keogh A, Lewis C, O'Connell J, Rogers J, Ross H, Russell S, Vanhaecke J; International Society of Heart and Lung Transplantation Guidelines. The International Society of Heart and Lung Transplantation Guidelines for the care of heart transplant recipients. J Heart Lung Transplant. 2010 Aug;29(8):914-56. doi: 10.1016/j.healun.2010.05.034. No abstract available. PMID 20643330
- [Background] Lund LH, Edwards LB, Kucheryavaya AY, Benden C, Dipchand AI, Goldfarb S, Levvey BJ, Meiser B, Rossano JW, Yusen RD, Stehlik J. The Registry of the International Society for Heart and Lung Transplantation: Thirty-second Official Adult Heart Transplantation Report--2015; Focus Theme: Early Graft Failure. J Heart Lung Transplant. 2015 Oct;34(10):1244-54. doi: 10.1016/j.healun.2015.08.003. Epub 2015 Aug 28. No abstract available. PMID 26454738